CLINICAL TRIAL: NCT00002951
Title: Hyperfractionated Radiotherapy With Concomitant Fluorouracil and Hydroxurea for Intermediate Stage Cancer of the Head and Neck
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8176; UCCRC-8176; NU-V96N1; NCI-G97-1159
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Esophageal Cancer; Head and Neck Cancer
Keywords: stage II esophageal cancer; stage III esophageal cancer; stage II nasopharyngeal cancer; stage III nasopharyngeal cancer; stage II lip and oral cavity cancer; stage III lip and oral cavity cancer; stage II hypopharyngeal cancer; stage III hypopharyngeal cancer; stage II laryngeal cancer; stage III laryngeal cancer; stage II paranasal sinus and nasal cavity cancer; stage III paranasal sinus and nasal cavity cancer; stage II oropharyngeal cancer; stage III oropharyngeal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Head and Neck Neoplasms; Nasopharyngeal Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms | interventions — Fluorouracil; Hydroxyurea; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Hyper-FHX) (Experimental): Concomitant chemoradiotherapy consisting of hydroxyurea (PO, BID, x 6days), continuous infusion 5-fluorouracil (IV, x 5days), hyperfractionated radiotherapy (150 cGy twice daily for 5 days every 14 days, 5 cycles)
  Interventions: Drug: fluorouracil; Drug: hydroxyurea; Procedure: surgical procedure; Radiation: radiation therapy

INTERVENTIONS:
Drug: fluorouracil
Drug: hydroxyurea
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy plus radiation therapy in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the locoregional control rates, time to failure, need for salvage surgery and overall survival of patients with intermediate stage cancer of the oral cavity, pharynx, larynx, paranasal sinuses, and cervical esophagus.
* Measure the impact of concomitant Hyper-FHX radiotherapy on organ preservation, organ function and quality of life parameters.
* Identify possible prognostic factors for toxic effects and response by performing pharmacologic monitoring.

OUTLINE: Patients receive concomitant chemoradiotherapy with curative intent. Patients who have microscopic or macroscopic residual disease 6 weeks after completion of chemoradiotherapy will receive a surgical salvage procedure.

The first cycle of chemotherapy will begin with PO doses of hydroxyurea every 12 hours on days 0-5. Fluorouracil is given IV on days 0-4. Radiation therapy BID is given on days 1-6. Cycles repeat every 14 days for a total of 5 cycles.

The disease will be reevaluated 4-6 weeks after completion of all treatment, every 3 months for 1 year, then yearly.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of carcinoma
* Stage II-III (T2, T3, N0 or T1-3, N1) carcinoma of head and neck, including: oral cavity, pharynx, larynx, paranasal sinuses, and cervical esophagus
* No N2 or N3
* Measurable disease is not required

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-3

Life expectancy:

* Anticipated survival is 3-4 years (median)

Hematopoietic:

* WBC count at least 3.5/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* Not specified

Pulmonary:

* Not specified

Other:

* No infection or severe medical illness
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* No prior surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 1996-06; Primary Completion 2004-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Locoregional control rate | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Everett E. Vokes, MD, Study Chair — University of Chicago
Locations (4):
- United States (4):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois

REFERENCES:
- [Result] Cohen EE, Haraf DJ, List MA, Kocherginsky M, Mittal BB, Rosen F, Brockstein B, Williams R, Witt ME, Stenson KM, Kies MS, Vokes EE. High survival and organ function rates after primary chemoradiotherapy for intermediate-stage squamous cell carcinoma of the head and neck treated in a multicenter phase II trial. J Clin Oncol. 2006 Jul 20;24(21):3438-44. doi: 10.1200/JCO.2006.05.8529. PMID 16849759